CLINICAL TRIAL: NCT04402541
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetic Profiles of CB-5339 in Participants With Relapsed/Refractory Acute Myeloid Leukemia or Relapsed/Refractory Intermediate or High Risk Myelodysplastic Syndrome
Brief Title: Study of CB-5339 in Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cleave Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTX-001
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CB-5339 (Experimental): Orally administered CB-5339
  Interventions: Drug: CB-5339

INTERVENTIONS:
Drug: CB-5339 — 25mg and 75mg capsules
  Other Names: CB-5339 Tosylate

SUMMARY:
This is a multicenter, open-label Phase 1 study of orally administered CB-5339 in participants with R/R AML or participants with R/R intermediate- to high-risk MDS.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1 study of orally administered CB-5339 in participants with R/R AML or participants with R/R intermediate- to high-risk MDS. The study will include two parts:1) a Dose Escalation phase in participants with R/R AML, or R/R intermediate- to high-risk MDS and 2) a Dose Expansion phase in participants with R/R AML for whom there is no standard of care therapy available that is likely to lead to disease remission. Additional cohorts for participants with R/R intermediate- to high-risk MDS following hypomethylating agents or other AML cohorts may be added at a later time.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and ≥ 18 years of age at the time of signing the consent form
2. One of the following advanced hematologic malignancies including:

   * Relapsed or refractory AML as defined by 2016 WHO criteria and are not candidates for curative therapies such as allogeneic hematopoietic cell transplant or for whom there is no standard of care therapy available that is likely to lead to disease remission according the investigator
   * MDS high-very high risk by the revised international scoring system for evaluating prognosis in myelodysplastic syndromes that is recurrent or refractory or the participant is intolerant to established therapy known to provide clinical benefit for their condition (e.g., relapsed following treatment with hypomethylating agent or lack of response after > 4 cycles), according to treating physician. Potential participants who meet the criteria for intermediate risk may be considered with approval by the medical monitor if the participant has severe cytopenia(s) and/or elevated bone marrow blast counts.
3. Adequate organ function defined as:

   * Serum creatinine ≤1.5 mg/dL or an estimated glomerular filtration rate of ≥60 mL/min as calculated by the Cockcroft-Gault glomerular filtration rate equation
   * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN) unless considered due to Gilbert's disease or leukemic disease
   * Aspartate aminotransferase (AST) ≤3 × the ULN; alanine aminotransferase (ALT) ≤3 × the ULN. Levels of AST and/or ALT ≤5 × the ULN may be acceptable for participants with known leukemic involvement of the liver after discussion with the study medical monitor
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
5. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If of childbearing potential, agree to use an effective barrier method of birth control (i.e., latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy during the study and 90 days after the last dose of CB-5339. Female participants of childbearing potential need a negative serum or urine pregnancy test within 7 days of study enrollment. Non-childbearing is defined as ≥ 1 year postmenopausal or surgically sterilized
6. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

1. Acute promyelocytic leukemia with t(15;17)(q22;q12); or abnormal promyelocytic leukemia/retinoic acid receptor alpha (PML-RARA).
2. Participants with clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid is only required if there is a clinical suspicion of CNS involvement by leukemia during screening.
3. Participants with immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
4. Concomitant malignancy, requiring active treatment, except for basal-cell or squamous cell carcinoma of the skin, carcinoma-in-situ of the uterine cervix, or localized prostate cancer.

   • Adjuvant therapy for breast cancer or prostate cancer is allowed.
5. Active, uncontrolled, systemic infection or severe localized infection during screening or prior to Cycle 1 Day 1 (C1D1; unless considered due to tumor by the investigator).

   • Note, participants receiving prophylactic anti-infectives are allowed on study.
6. Known human immunodeficiency virus (HIV) infection with CD4+ T cell counts <350 cells/μL, initiation of antiretroviral therapy within 4 weeks before C1D1, or acquired immunodeficiency syndrome (AIDS)-related infection within 12 months before C1D1.
7. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with viral load above the limit of quantification
8. Major cardiac abnormalities as defined but not limited to the following: uncontrolled angina or unstable life-threatening arrhythmias, history of myocardial infarction within 12 weeks prior to Baseline, Class 3 or higher New York Heart Association (NYHA) congestive heart failure, or left ventricular ejection fraction (LVEF) <45% as measured by echocardiogram (ECHO) within 28 days of C1D1
9. Persistent (3 consecutive ECGs performed ≥5 minutes apart) prolongation of the corrected QT interval by Fredericia's method (QTcF) to > 480 msec
10. Gastrointestinal conditions that may interfere with the absorption of orally-administered drugs including but not limited to short gut syndrome, gastroparesis, inflammatory bowel disease, or acute pancreatitis.
11. Any other severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or CB-5339 administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, may interfere with the interpretation of the study results and, in the Investigator's opinion, or would make the participant inappropriate for entry into this study
12. A condition that is expected to require concomitant use of any medication listed as prohibited while on study.
13. Known hypersensitivity to any components of CB-5339.
14. Use of chemotherapy (except hydroxyurea), radiation or monoclonal antibodies within 14 days or 5 half-lives for small molecule inhibitors prior to first dose of CB-5339
15. Participants who have undergone a hematopoietic cell transplant (HCT) within 100 days of the first dose of CB-5339, or participants on immunosuppressive therapy post-HCT at the time of screening, use of calcineurin inhibitors within 4 weeks prior to first dose of CB-5339, or with clinically significant graft-versus-host disease (GVHD).

    • Note: The use of topical steroids or <10mg oral prednisone for ongoing skin GVHD is permitted.
16. Major surgery within 4 weeks prior to first dose of CB-5339. Participant must have recovered from surgery and be without current complications of infection or dehiscence
17. Enrollment in other clinical trials unless approved by Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-07-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | 28 Days
Define the MTD and/or RP2D and schedule for CB-5339 | 28 Days
  Incidence and nature of DLTs with CB-5339 monotherapy for MTD determination. All available safety, efficacy and PK, for RP2D determination

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Day 1 and Day 4
Time to reach peak plasma concentration (Tmax) | Day 1 and Day 4
Area under the plasma concentration time curve (AUC0-t) | Day 1 and Day 4
Elimination half-life (t½) | Day 1 and Day 4
Accumulation ratio | Day 1 and Day 4
Antitumor effects | End of each cycle (cycle is 28 days)
  CR/CRi rate at the RP2D in participants with R/R AML, as assessed by the investigator, based on 2017 ELN response criteria.
  Objective response rate (ORR) at the RP2D in participants with R/R AML, as assessed by the investigator based on 2017 ELN response criteria.
  DoCR in participants with R/R AML who attain CR or CRi

CONTACTS AND LOCATIONS:
Overall Officials: Scott Harris, Study Chair — Cleave Therapeutics, Inc.
Locations (10):
- United States (7):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - KU Clinical Research Center, Fairway, Kansas
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornel Medical Center, New York, New York
  - Saint Francis Hospital Cancer Center, Greenville, North Carolina
  - Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MD Anderson Cancer Cancer, Houston, Texas
- Australia (3):
  - St. Vincent Hospital, Sydney, NSW, Darlinghurst, New South Wales
  - Epworth Healthcare, Melbourne, Victoria
  - Haematology Clinical Trials Unit, Royal Perth Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Wang F, Li S, Rosencrans WM, Cheng KW, Stott GM, Mroczkowski B, Chou TF. Sulforaphane is Synergistic with CB-5083 and Inhibits Colony Formation of CB-5083-Resistant HCT116 Cells. ChemMedChem. 2022 Jun 3;17(11):e202200030. doi: 10.1002/cmdc.202200030. Epub 2022 Apr 22. PMID 35451199